CLINICAL TRIAL: NCT03555305
Title: Relative Bioavailability of LY2963016 to LANTUS® After Single-Dose Subcutaneous Administration in Healthy Chinese Subjects
Brief Title: A Study of Insulin Glargine (LY2963016) in Healthy Chinese Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 13877; I4L-MC-ABEF (Other: Eli Lilly and Company)
Record Dates: First submitted 2018-06-01; First posted 2018-06-13 (Actual); Results first posted 2020-11-24 (Actual); Last update posted 2020-11-24 (Actual); Status verified 2019-11-15

CONDITIONS: Healthy
MeSH Terms: interventions — Insulin Glargine; LY2963016 insulin glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Insulin Glargine (Experimental): Participants received 0.5 units per kilogram (U/kg) of Insulin Glargine subcutaneously (SC).
  Interventions: Drug: Insulin Glargine
- Lantus (Active Comparator): Participants received 0.5 U/Kg of Lantus subcutaneously.
  Interventions: Drug: Lantus

INTERVENTIONS:
Drug: Insulin Glargine — Administered SC
  Other Names: LY2963016; Basaglar
  Arms: Insulin Glargine
Drug: Lantus — Administered SC
  Other Names: Insulin Glargine
  Arms: Lantus

SUMMARY:
The purpose of this study is to compare a study drug known as Insulin glargine with Lantus in healthy Chinese participants. Blood samples will be taken to compare how the body handles the drugs and how they affect blood sugar levels. Side effects and tolerability will be documented. The study will last at least 18 days, not including screening. Screening is required within 4 weeks prior to the start of the study.

ELIGIBILITY:
Inclusion Criteria:

* Are native Chinese men or women. Native Chinese is defined as a participant who has both parents and all 4 grandparents of Chinese origin.
* For females of childbearing potential (defined as not surgically sterilised and between menarche and 1-year postmenopause) only:

  * Negative serum pregnancy test at the time of screening.
  * Are not lactating.
  * Intend not to become pregnant during the study.
  * Are sexually inactive or have practiced a reliable method of birth control for at least 6 weeks prior to screening.
  * Agree to continue to use a reliable method of birth control (as determined by the investigator) during the study.
* For females not of childbearing potential, must be:

  * Surgically sterile, defined as having had a hysterectomy or bilateral oophorectomy or tubal ligation, and/or
  * Menopausal, defined as having had no menses for at least 1 year, or a plasma follicular stimulating hormone value of >40 milli-international units per milliliter (mIU/mL) and no menses for at least 6 months, unless the participant is taking hormone-replacement therapy.
* Having fasting plasma glucose <110 milligrams per deciliter (mg/dL) (<6.1 millimoles per liter [mmol/L]) and 2-hour glucose level <140 mg/dL (<7.8 mmol/L) on the 75 grams (g) oral glucose tolerance test.
* Have a body mass index (BMI) between 18 and 28 kilograms per meter squared (kg/m²), inclusive, at screening.
* Are nonsmokers, have not smoked for at least 6 months prior to entering the study, and agree not to smoke (cigars, cigarettes, or pipes) or use smokeless tobacco for the duration of the study.
* Have normal blood pressure and pulse rate at screening, as determined by the investigator.
* Have an electrocardiogram (ECG), at screening, considered as within normal limits by the investigator.
* Have clinical laboratory test results within normal reference range for the population or investigator site, or results with acceptable deviations that are judged to be not clinically significant by the investigator.

Exclusion Criteria:

* Have a history of first-degree relatives known to have diabetes mellitus.
* Have known allergies to insulin glargine or its excipients, or related drugs, or heparin, or have a history of relevant allergic reactions of any origin.
* Have a significant history of or current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, haematological, or neurological disorders capable of significantly altering the absorption, metabolism, or elimination of drugs; of constituting a risk when taking the study medication; or of interfering with the interpretation of data.
* Show evidence of human immunodeficiency virus infection (HIV) and/or positive human HIV antibodies.
* Have positive hepatitis B surface antigen.
* Have donated >400 mL of blood in the last 6 months or donated >100 mL within the last 30 days.
* Have an average weekly alcohol intake that exceeds 21 units per week (males) and 14 units per week (females), or are unwilling to stop alcohol consumption while resident in the clinical research unit (CRU) (1 unit = 12 ounces or 360 mL of beer; 5 ounces or 150 mL of wine; 1.5 ounces or 45 mL of distilled spirits).
* Intend to use: prescription medication or over-the-counter medication or Chinese traditional medicine within 14 days before dosing (apart from vitamin/mineral supplements, occasional paracetamol, thyroid replacement, or birth control methods). If this situation arises, an otherwise suitable participant may be included at the discretion of the investigator.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2019-11-04 (Actual); Study Completion 2019-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Liu H, Wang F, Ji Y, Ma T, Li H, Linnebjerg H, Chua L, Tham LS, Yu Y. A Euglycemic Glucose Clamp Study to Evaluate the Bioavailability of LY2963016 Relative to Insulin Glargine in Healthy Chinese Subjects. Clin Pharmacol Drug Dev. 2021 Dec;10(12):1452-1459. doi: 10.1002/cpdd.1014. Epub 2021 Aug 19. PMID 34410042

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two period crossover study, with a minimum of 7 days washout period between each period.
Groups:
- Sequence 1: Period 1: Participants received 0.5 units per kilogram (U/kg) of Insulin glargine subcutaneously.
  Period 2: Participants received 0.5 U/Kg of Lantus subcutaneously.
- Sequence 2: Period 1: Participants received 0.5 U/Kg of Lantus subcutaneously. Period 2: Participants received 0.5 U/Kg of Insulin glargine subcutaneously.
Period: Period 1
Arm/Group | Sequence 1 | Sequence 2
Started | 29 | 29
Received at Least 1 Dose of Study Drug | 29 | 29
Completed | 29 | 27
Not Completed | 0 | 2
Not completed — Physician Decision | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Period 2
Arm/Group | Sequence 1 | Sequence 2
Started | 29 | 27
Completed | 29 | 27
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study drug.
Groups:
- Overall: Participants received 0.5 U/Kg of Insulin glargine and Lantus subcutaneously as per dosing schedule.
Arm/Group | Overall
Number analyzed (Participants) | 58
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.9 (2.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 58
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 58
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  China | 58

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics (PK): Maximum Serum Concentration (Cmax) of Insulin Glargine and Lantus
Description: Pharmacokinetics (PK): Maximum Serum Concentration (Cmax) of Insulin glargine and Lantus.
Time Frame: -0.5 and 0 hours predose; 0.5, 1, 2, 3, 4, 6, 9, 12, 15, 18, 21, and 24 hours postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole per liter (pmol/L)
Groups:
- 0.5 U/kg Insulin Glargine: Participants received single 0.5 U/kg dose of Insulin glargine administered subcutaneously.
- 0.5 U/kg Lantus: Participants received single 0.5 U/kg dose of Lantus administered subcutaneously.
Arm/Group | 0.5 U/kg Insulin Glargine | 0.5 U/kg Lantus
Number analyzed (Participants) | 56 | 58
picomole per liter (pmol/L) | 124 (31) | 129 (33)
Statistical Analysis 1: Comparison: 0.5 U/kg Insulin Glargine vs 0.5 U/kg Lantus; Test type: Equivalence — Analysis was performed using linear mixed effects model and participant as a random effect, with period, sequence, and treatment as fixed effects. The estimate of the ratio of means of each PK/PD parameters between the 2 treatments and the corresponding 90% confidence interval were calculated. A typical bio-equivalence limit (0.8 to 1.25) was used as equivalence margin; Linear mixed-effects model; Ratio of geometric least squares means = 0.961, 90% CI 2-sided [0.886 to 1.04]

2. Primary Outcome: PK: Area Under the Concentration Versus Time Curve From Time Zero to 24 Hours (AUC[0-24]) of Insulin Glargine and Lantus
Description: PK: Area Under the Concentration Versus Time Curve From Time Zero to 24 Hours (AUC[0-24]) of Insulin glargine and Lantus.
Time Frame: -0.5 and 0 hours predose; 0.5, 1, 2, 3, 4, 6, 9, 12, 15, 18, 21, and 24 hours postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable PK data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picomole*hour per liter (pmol*hr/L)
Arm/Group | 0.5 U/kg Insulin Glargine | 0.5 U/kg Lantus
Number analyzed (Participants) | 56 | 58
picomole*hour per liter (pmol*hr/L) | 2170 (28) | 2310 (29)
Statistical Analysis 1: Comparison: 0.5 U/kg Insulin Glargine vs 0.5 U/kg Lantus; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Linear mixed-effects model; Ratio of geometric least squares means = 0.943, 90% CI 2-sided [0.874 to 1.02]

3. Secondary Outcome: Pharmacodynamics (PD): Total Amount of Glucose Infused (Gtot)
Description: Gtot was the total glucose infusion over the clamp duration and was used to measure the study drug action over time as measured by the euglycaemic clamp procedure. During the euglycaemic clamp procedure, blood glucose concentrations were held constant after the administration of Insulin glargine or Lantus by adjusting the exogenous glucose infusion rate. Data presented were adjusted by the body weight.
Time Frame: 30 minutes predose through 24 hours postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable Gtot data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams/kilogram (mg/kg)
Arm/Group | 0.5 U/kg Insulin Glargine | 0.5 U/kg Lantus
Number analyzed (Participants) | 56 | 58
milligrams/kilogram (mg/kg) | 2390 (43) | 2680 (40)

4. Secondary Outcome: PD: Maximum Glucose Infusion Rate (Rmax)
Description: Rmax is the maximum infusion rate of glucose administered intravenously needed to maintain target blood glucose level and is used to measure the study drug action over time as measured by the euglycaemic clamp procedure. During the euglycaemic clamp procedure, blood glucose concentrations are held constant after the administration of Insulin glargine or Lantus by adjusting the exogenous glucose infusion rate. Data presented were adjusted by the body weight.
Time Frame: 30 minutes predose through 24 hours postdose
Population: All randomized participants who received at least one dose of study drug and had evaluable Rmax data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: milligrams/kilograms/minute (mg/kg/min)
Arm/Group | 0.5 U/kg Insulin Glargine | 0.5 U/kg Lantus
Number analyzed (Participants) | 56 | 58
milligrams/kilograms/minute (mg/kg/min) | 2.72 (37) | 2.99 (36)

ADVERSE EVENTS:
Time Frame: Up to 14 Days
Description: All randomized participants who received at least one dose of study drug.
Arm/Group | 0.5 U/kg Insulin Glargine | 0.5 U/kg Lantus
All-Cause Mortality (participants affected / at risk) | 0/56 | 0/58
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/58
Other Adverse Events (participants affected / at risk) | 0/56 | 0/58

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/05/NCT03555305/Prot_000.pdf
  • Statistical Analysis Plan (2019-05-06): https://cdn.clinicaltrials.gov/large-docs/05/NCT03555305/SAP_001.pdf